CLINICAL TRIAL: NCT01551043
Title: Pilot Study of Donor Lymphocyte Infusions Using Donor T Cells Engineered to Contain Anti-CD19 Attached To TCR And 4-1BB Signaling Domains in Patients With Relapsed CD19+ All After Allogeneic Stem Cell Transplantation
Brief Title: Allo CART-19 Protocol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative Reasons
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01410
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: adult patients; aged 18; CD19+ ALL relapsed; after allogeneic SCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19

SUMMARY:
The primary objective is to determine the safety and survival of the redirected allogeneic T cells transduced with the anti-CD19 lentiviral vector (referred to as CART-19 cells).

DETAILED DESCRIPTION:
The investigators propose an open label, single center, pilot study to evaluate the safety and tolerability, and persistence of donor lymphocytes engineered to express a chimeric antigen receptor targeting CD19 which is linked to the CD3:4-1BB signaling chains in patients with CD19+ acute lymphoblastic leukemia (ALL). Upon enrollment, donors will undergo leukapheresis and patients will undergo an optional bone marrow/lymph node biopsy approximately four weeks prior to dosing. Between dosing and treatment, patients may undergo an additional chemotherapy treatment depending upon their disease. At dosing, patients will receive redirected donor lymphocytes targeted against CD19 (allo-CART-19 cells). The cell dose will be given as a split infusion over three days to enhance the ability to manage any infusion related toxicity. Patients will be monitored weekly for four weeks. At the end of four weeks, patients will undergo a second leukapheresis and second optional bone marrow/lymph node biopsy. At this point the patient will also undergo restaging. Observation and monitoring of patients will continue on a monthly basis until week 24 post dosing. Annual follow-up for lentiviral vector safety will be carried out for 15 years in accordance with FDA guidelines for retroviral vectors. Ten subjects will be targeted for this study, with an expected rate of drop out of 30% due to disease progression between enrollment and week four post dosing.

ELIGIBILITY:
Inclusion Criteria:

* CD19+ ALL relapsed after allogeneic SCT.
* No active GVHD and off immunosuppression for greater than or equal to 4 weeks.
* Age greater than or equal to 18 years.
* Creatinine less than or equal to2.5 mg/dl.
* ALT/AST less than or equal to3x normal
* Bilirubin less than or equal to2.0 mg/dl
* Donor is available and is able to undergo apheresis. A separate donor consent process and form is described below.
* Voluntary informed consent is given.

Exclusion Criteria:

* Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene therapy products.
* Feasibility assessment during screening demonstrates less than 30% transduction of target lymphocytes, or insufficient expansion ( less than 5-fold) in response to CD3/CD28 costimulation..
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* HIV infection.
* Patients with active CNS involvement with leukemia. Patients with prior CNS disease that has been effectively treated will be eligible providing treatment was greater than or equal to 4 weeks before enrollment
* Patients with active GVHD or requiring immune suppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States